CLINICAL TRIAL: NCT03690921
Title: Linear Energy Transfer (LET)-Optimized Intensity Modulated Proton Therapy (IMPT) as a Component of Definitive Chemoradiation for Newly Diagnosed Squamous Cell Carcinoma of the Anal Canal: a Feasibility Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0420; NCI-2018-02040 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0420 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anal Canal Squamous Cell Carcinoma; Stage I Anal Cancer AJCC v8; Stage II Anal Cancer AJCC v8; Stage IIA Anal Cancer AJCC v8; Stage IIB Anal Cancer AJCC v8; Stage III Anal Cancer AJCC v8; Stage IIIA Anal Cancer AJCC v8; Stage IIIB Anal Cancer AJCC v8; Stage IIIC Anal Cancer AJCC v8
MeSH Terms: conditions — Anus Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorouracil; dehydroftorafur; Linear Energy Transfer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (LET-IMPT, chemotherapy) (Experimental): Patients undergo linear energy transfer-optimized intensity modulated proton therapy 5 times per week for 5-6 weeks. Patients also receive standard cisplatin and fluorouracil IV weekly for up to 6 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Fluorouracil; Radiation: Linear Energy Transfer-Optimized Intensity Modulated Proton Therapy; Procedure: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Radiation: Linear Energy Transfer-Optimized Intensity Modulated Proton Therapy — Undergo LET-IMPT
  Other Names: LET-Optimized IMPT; LET-Optimized Intensity Modulated Proton Therapy; Linear Energy Transfer (LET)-Optimized Intensity Modulated Proton Therapy (IMPT)
Procedure: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the side effects of LET-IMPT and standard chemotherapy, and how well they work in treating patients with newly diagnosed stage I-III anal canal squamous cell cancer. LET-IMPT is a type of radiation therapy that uses high energy proton "beamlets" to "paint" the radiation dose into the target and may help to kill tumor cells and shrink tumors. Giving LET-IMPT and standard chemotherapy may work better in treating patients with anal canal squamous cell cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess physician-reported acute grade 3 or greater gastrointestinal, genitourinary and hematologic toxicities at 12 weeks post-treatment for patients treated with linear energy transfer (LET)-optimized, intensity-modulated proton therapy (IMPT) and compare to contemporary controls treated with volume modulated arc therapy (VMAT) to determine the feasibility of this outcome for a future randomized trial.

SECONDARY OBJECTIVES:

I. To assess the feasibility of enrolling patients on a prospective trial delivering LET-optimized IMPT for newly diagnosed, non-metastatic anal cancer.

II. To develop guidelines and workflow to create and deliver anal canal cancer treatments using LET-optimized IMPT.

III. To evaluate complete response rate at 12 weeks and 24 weeks post-treatment.

IV. To evaluate local progression free survival, distant metastasis-free survival and overall survival at 24 and 48 months.

V. To evaluate rates of patient-reported acute toxicity, function, distress and quality of life (QOL) at 12 weeks.

VI. To evaluate rates of patient-reported late toxicity, function, distress and QOL every 6 months for 24 months.

VII. To evaluate the value of proton therapy by comparing Time-Driven Activity-Based Costing data from the date of consultation until the date of the 12-week follow up visit post-treatment with contemporary controls treated with VMAT.

EXPLORATORY OBJECTIVES:

I. To compare dose to the pelvic bone marrow, bowel, bladder and genitalia between LET-optimized IMPT, traditionally-optimized IMPT and VMAT.

II. To assess rates of leukopenia, neutropenia and lymphopenia at 12-weeks post-treatment for patients treated with LET-optimized IMPT and compare to contemporary controls treated with VMAT.

III. To correlate white blood cell counts (WBC), absolute neutrophil counts (ANC) and absolute lymphocyte counts (ALC) with dose to the pelvic bone marrow for patients treated with LET-optimized IMPT.

OUTLINE:

Patients undergo linear energy transfer-optimized intensity modulated proton therapy 5 times per week for 5-6 weeks. Patients also receive standard cisplatin and fluorouracil intravenously (IV) weekly for up to 6 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven, non-metastatic invasive primary squamous cell carcinoma of the anal canal (stages I, II, and III)
* History/physical examination including documentation of the primary anal lesion size, distance from the anal verge and anal sphincter tone within 60 days prior to registration
* Anal examination with biopsy on either colonoscopy, sigmoidoscopy, rigid proctoscopy or anoscopy
* Computed tomography (CT) scan of the chest and abdomen with contrast or contrast-enhanced positron emission tomography (PET)/CT scan within 60 days of registration unless the patient has a documented contrast allergy
* CT scan of pelvis with contrast or contrast-enhanced PET/CT scan within 60 days of registration unless the patient has a documented contrast allergy
* Zubrod performance status of 0-1 within 60 days prior to registration
* Absolute neutrophil count (ANC) >=1.8 K/ul, cannot be achieved through granulocyte-colony stimulating factor (GCSF) (within 30 days prior to study registration)
* Platelets >= 100 K/uL, cannot be achieved through transfusion (within 30 days prior to study registration)
* Hemoglobin >= 8 g/dL, cannot be achieved through transfusion (within 30 days prior to study registration)
* Serum creatinine =< 1.5 mg/dL (within 30 days prior to study registration)
* Bilirubin =< 1.4 mg/dL, except in the case of patients with Gilbert's disease (within 30 days prior to study registration)
* White blood cells (WBC) >= 3000/microliter (within 30 days prior to study registration)
* Aspartate transaminase (AST)/alanine transaminase (ALT) < 3 x the upper limit of normal (within 30 days prior to study registration)
* International normalized ratio (INR) =< 1.5 (within 30 days prior to study registration)
* Human Immunodeficiency Virus (HIV) test must be done within 30 days of study registration. If HIV positive, CD4 count must be obtained within 30 days of study registration

  * Note: HIV positive patients are eligible for this study if they have a CD4 count > 400 cells/mm^3
* The patient must either have insurance authorization or otherwise secure funding to cover IMPT
* The patient must be able to receive concurrent chemotherapy

Exclusion Criteria:

* Prior invasive malignancy (except non-melanomatous skin cancer), unless disease free for a minimum of 3 years
* Prior systemic chemotherapy for anal cancer
* Prior radiotherapy to the pelvis that would result in overlap of radiation fields
* Evidence of distant metastatic disease (M1)
* Prior surgery to the anal canal that removed all macroscopic anal cancer
* Women of childbearing potential or men who do not agree to use a medically effective form of birth control throughout their participation in the treatment phase of the study
* Severe, active co-morbidity defined as follows: unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; transmural myocardial infarction within the last 6 months; acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; HIV positive with a CD4 count < 400 cells/mm^3; other immuno-compromised status; women who are pregnant or lactating; uncontrolled infection as deemed by the principal investigator (PI); patient incarceration

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma B Holliday, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from 11/5/2018 until 6/3/2022. Recruitment occurred in radiation oncology clinics at UT MD Anderson Cancer Center.
Pre-assignment Details: There were no enrolled patients excluded prior to assignment to arms or groups.
Groups:
- IMPT for Anal Cancer (Single Arm Trial): Intensity Modulated Proton Therapy with concurrent chemotherapy as definitive treatment for non-metastatic anal squamous cell carcinoma.
Period: Overall Study
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 70 [68.5 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Acute Toxicity
Description: Number (percentage) of patients with physician-reported acute G3+ GI, GU and heme toxicities
Time Frame: Acute physician reported toxicity from start of treatment 12 weeks post-treatment
Population: All patients with 12 week follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 2

2. Secondary Outcome: Complete Response at 12 Weeks
Description: Number (percentage) patients who achieved a complete clinical response of their disease by 12 weeks after chemoradiation.
Time Frame: 12 weeks
Population: All patients with 12 weeks follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 6

3. Secondary Outcome: Local Progression Free Survival at 24 Months
Description: Patients alive without evidence of local progression 24 months after chemoradiation.
Time Frame: 24 months
Population: Patients with 24 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 5

4. Secondary Outcome: Distant Metastasis-free Survival at 24 Months.
Description: Patients alive without evidence of distant metastases 24 months after chemoradiation.
Time Frame: 24 months
Population: Patients with 24 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 5

5. Secondary Outcome: Overall Survival at 24 Months
Description: Patients alive 24 months after chemoradiation.
Time Frame: 24 months
Population: Patients with 24 month follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 7

6. Secondary Outcome: Complete Response at 24 Weeks
Description: Number (percentage) patients who achieved a complete clinical response of their disease by 24 weeks after chemoradiation.
Time Frame: 24 weeks
Population: All patients with 24 week follow up
Measure: Count of Participants; unit: Participants
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
Number analyzed (Participants) | 8
Participants | 6

ADVERSE EVENTS:
Time Frame: Assessed up to 2 years
Description: CTCAE v4
Groups:
- IMPT for Anal Cancer (Single Arm Trial): Acute physician reported toxicity from start of treatment 12 weeks post-treatment.
Arm/Group | IMPT for Anal Cancer (Single Arm Trial)
All-Cause Mortality (participants affected / at risk) | 1/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMPT for Anal Cancer (Single Arm Trial) (N=8)
Abnormal bowel habits (Gastrointestinal disorders) | 1 (1)
Absolute eosinophil decrease (Blood and lymphatic system disorders) | 3 (3)
Absolute lymphocyte decrease (Blood and lymphatic system disorders) | 5 (5) — Grade 1
Absolute lymphocyte decrease (Blood and lymphatic system disorders) | 7 (7) — Grade 2
Absolute lymphocyte decrease (Blood and lymphatic system disorders) | 7 (7) — Grade 3
Absolute lymphocyte decrease (Blood and lymphatic system disorders) | 1 (1) — Grade 4 lymphopenia is numerically defined as a value less than 200 cells per microliter. It is not considered a serious medical event as it is not life-threatening, require hospitalization, intervention and does not impact delivery of treatment.
Absolute monocyte decrease (Blood and lymphatic system disorders) | 4 (4)
Absolute neutrophil decrease (Blood and lymphatic system disorders) | 2 (2)
Absolute neutrophil increase (Blood and lymphatic system disorders) | 2 (2) — Grade 1
Absolute neutrophil increase (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Acute kidney disease (Renal and urinary disorders) | 1 (1)
Alkaline phosphatase increase (Blood and lymphatic system disorders) | 1 (1) — Grade 1
Alkaline phosphatase increase (Blood and lymphatic system disorders) | 1 (1) — Grade 2
Anal fissure (Gastrointestinal disorders) | 1 (1)
Anal bleeding (Gastrointestinal disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 7 (7)
Anorectal pain (Gastrointestinal disorders) | 1 (1)
Anorectal pain (Gastrointestinal disorders) | 3 (3) — Grade 2
Anorexia (Gastrointestinal disorders) | 1 (1)
AST Increased (Blood and lymphatic system disorders) | 1 (1)
Back pain (Gastrointestinal disorders) | 1 (1)
Bilateral foot pain (Nervous system disorders) | 1 (1)
Binaural tinnitus (Nervous system disorders) | 1 (1)
Bladder incontinence (Renal and urinary disorders) | 1 (1)
Bowel incontinence (Gastrointestinal disorders) | 1 (1)
Bowel urgency (Gastrointestinal disorders) | 1 (1)
BUN increase (Renal and urinary disorders) | 3 (3)
Carbon Dioxide Decreased (Blood and lymphatic system disorders) | 1 (1)
Chest pain (non-cardiac) (Gastrointestinal disorders) | 1 (1)
Chloride level increase (Metabolism and nutrition disorders) | 1 (1)
Chloride level decrease (Metabolism and nutrition disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) — Grade 1
Constipation (Gastrointestinal disorders) | 2 (2) — Grade 2
Creatinine increased (Renal and urinary disorders) | 5 (5)
Dermatitis (Skin and subcutaneous tissue disorders) | 5 (5) — Grade 1
Dermatitis (Skin and subcutaneous tissue disorders) | 6 (6) — Grade 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3
Diarrhea (Gastrointestinal disorders) | 5 (5) — Grade 1
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 2
Diarrhea (Gastrointestinal disorders) | 1 (1) — Grade 3
Difficulty with sleep (General disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspaurenia (Skin and subcutaneous tissue disorders) | 1 (1)
Epigastric pain (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 5 (5) — Grade 1
Fatigue (General disorders) | 2 (2) — Grade 2
High TSH (Metabolism and nutrition disorders) | 1 (1)
Hot flashes (Metabolism and nutrition disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7) — Grade 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — Grade 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 5 (5) — Grade 1
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) — Grade 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) — Grade 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) — Grade 2
Increased LDH (Metabolism and nutrition disorders) | 1 (1)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 1
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Low TSH (Metabolism and nutrition disorders) | 1 (1)
Lower extremity edema (Musculoskeletal and connective tissue disorders) | 1 (1)
Maculopapular rash of torso (Skin and subcutaneous tissue disorders) | 1 (1)
Monocyte count increase (Blood and lymphatic system disorders) | 1 (1)
Mucous discharge (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (5)
Nosebleed (Blood and lymphatic system disorders) | 1 (1)
PICC line pain (General disorders) | 2 (2)
Platelet count decreased (Blood and lymphatic system disorders) | 2 (2)
Total protein decreased (Metabolism and nutrition disorders) | 3 (3)
Ear fullness (General disorders) | 1 (1)
Troponin I increased (Cardiac disorders) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (1)
Urinary Urgency (Renal and urinary disorders) | 1 (1)
White blood cell count decreased (Blood and lymphatic system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT03690921/Prot_SAP_001.pdf